CLINICAL TRIAL: NCT04874272
Title: Feasibility and Acceptability of a Chaplain-Led Post-Code Debrief Intervention
Acronym: PCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other); Daniel F. Evans Center for Spiritual and Religious Values in Healthcare (Unknown)
Responsible Party: Principal Investigator, Shelley E. Varner Perez, Senior Program Manager, Research Chaplain, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006053247
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Health Personnel Attitude

STUDY DESIGN:
Intervention Model Description: Phased single group study. Phase (arm) 1: Participants complete a survey Phase (arm) 2- Pilot (single hospital unit): Participants attend a chaplain led post-code debrief, complete a survey Phase (arm) 3 (multiple hospital units): Participants attend a chaplain led post-code debrief, complete a survey.
  During all phases participants may be approached to complete an additional interview with the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Intervention (No Intervention): Pre-intervention: participants complete research surveys about codes and are asked to participate in an interview with the research team.
- Pilot (Single Unit Recruitment) (Experimental): Pilot intervention: participants participate in a chaplain led post-code debrief, participants complete research surveys about codes.
  Interventions: Other: Chaplain led post-code debrief
- Pilot (Hospital-wide Recruitment) (Experimental): Pilot intervention: participants participate in a chaplain led post-code debrief, participants complete research surveys about codes.
  Interventions: Other: Chaplain led post-code debrief

INTERVENTIONS:
Other: Chaplain led post-code debrief — an emotional debrief (a discussion to process the emotional, existential impact of a medical code/cardiopulmonary arrest), which will be led by a chaplain
  Arms: Pilot (Hospital-wide Recruitment); Pilot (Single Unit Recruitment)

SUMMARY:
The objective of this study is to increase the frequency and effectiveness of post code debriefs by piloting a novel intervention tool and partnering clinicians with board certified chaplains trained to facilitate group processes. A post code debrief will involve two aspects: a technical debrief (a discussion to process the technical, procedural aspects of a medical code/cardiopulmonary arrest), which will be led by a clinician, and an emotional debrief (a discussion to process the emotional, existential impact of a medical code/cardiopulmonary arrest), which will be led by a chaplain.

DETAILED DESCRIPTION:
Technical debriefs already are a familiar part of practice; the novel portion of this study is the introduction of the chaplain-led portion of emotional debrief. Also novel is the combination of the technical and emotional debriefs. As part of the study debrief, participants are asked to be present for and engaged in the discussion reviewing the code event, though there is no expectation or requirement for providing verbal input. Data about the content of the code debrief and the interventions provided during the debrief will be recorded by the Code Blue Chaplain in REDCap. Data about participants will be self-reported in their REDCap survey responses.

Clinicians who participate in resuscitation attempts during cardio-pulmonary arrests (CPA) experience psychological, emotional, and moral distress, including feelings of anxiety, grief, and regret. These experiences directly impact feelings of burnout, which is a leading cause in staff turnover. While debriefing soon after the experience has been shown to increase positive coping and reduce acute stress, post code debriefs are rarely conducted. Current models rely on physicians to facilitate debriefs and do not provide a standard tool. Physicians often feel untrained and uneasy with this role. To address these findings, we seek to implement a standardized post-code debriefing process that is co-led by a clinician and a chaplain.

Specific Aim 1: Evaluate and describe current stress of clinical staff who participate in CPA events. During the first six months of the grant period, a staff chaplain will respond to all "Code Blues." The chaplain will recruit at least five clinical staff participants from at least two different disciplines to complete surveys one-week and six-weeks after the CPA event.

Specific Aim 2: Pilot intervention to debrief CPA experience. During the second six months of the grant period, the research team will pilot the new debrief tool on the Cardiac Medical Critical Care Unit (CMCC). The designated "Code Blue" Chaplain will respond to all code blues on CMCC. The Code Blue Chaplain will be responsible for establishing the time and location of the Post Code Debrief, providing the technical debrief tool to a qualified clinician, and facilitating the emotional debrief following the semi-structured debrief tool. The Code Blue Chaplain will recruit participants to complete follow up surveys one-week and six-weeks following the CPA event.

Specific Aim 3: Assess feasibility and acceptability. Describe team member experience. During the final year of the grant period, the research team will expand the intervention tool throughout IU Health Methodist Hospital. The Code Blue Chaplain will respond to all overhead code blue pages and proceed with the intervention and recruiting as stated above.

ELIGIBILITY:
Inclusion Criteria for EVENT:

* Code event occurs on an adult inpatient unit at IU Health Methodist Hospital
* Cardiopulmonary arrest where cardiopulmonary resuscitation (CPR) was performed for at least one minute
* Code event occurs when at least two chaplains are available in the hospital.
* Patient involved is an inpatient
* Patient involved is over the age of 18
* Code is called on the overhead paging system

Inclusion Criteria for STAFF:

* Employee of participating hospital site
* Actively involved in the CPA in one of the following capacities:
* Gave compressions
* Administered medication
* Provided respiratory support
* Gave clinical orders or directions to staff
* Documented interventions during CPA
* Proficient in written and spoken English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Evaluate and describe current stress of clinical staff who participate in CPA events | 6 weeks
  Participants complete surveys at 1 and 6 weeks post-CPA event
Pilot the debrief tool on one unit of the hospital | 6 weeks
  Participants participate in the intervention (debrief) and complete surveys at 1 and 6 weeks post-CPA event
Pilot the debrief tool hospital-wide | 6 weeks
  Participants participate in the intervention (debrief) and complete surveys at 1 and 6 weeks post-CPA event

CONTACTS AND LOCATIONS:
Overall Officials: Shelley E Varner Perez, MDiv, MPH, Principal Investigator — Indiana University
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No